CLINICAL TRIAL: NCT05564338
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study to Compare the Efficacy and Safety of Sitravatinib Plus Tislelizumab or Placebo Plus Tislelizumab Versus Placebo as Adjuvant Treatment in Patients With Hepatocellular Carcinoma Who Are at High Risk of Recurrence After Surgical Resection
Brief Title: Efficacy and Safety of Sitravatinib Plus Tislelizumab or Placebo Plus Tislelizumab Versus Placebo as Adjuvant Treatment in Participants With Hepatocellular Carcinoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study has voluntarily discontinued due to a change in the company-level development strategy and is not because of any safety concern or the request from any health authority worldwide.
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGB-A317-Sitravatinib-303
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; sitravatinib; tislelizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sitravatinib; tislelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Arm A: sitravatinib + tislelizumab (Experimental): sitravatinib once daily and tislelizumab once every 6 weeks, for up to 17 cycles (approximately 2 years)
  Interventions: Drug: Sitravatinib; Drug: Tislelizumab
- Treatment Arm B: Placebo + tislelizumab (Experimental): sitravatinib-matching placebo once daily and tislelizumab once every 6 weeks, for up to 17 cycles (approximately 2 years)
  Interventions: Drug: Tislelizumab; Drug: sitravatinib-matching placebo
- Treatment Arm C:Sitravatinib + Placebo (Experimental): sitravatinib once daily and tislelizumab-matching placebo once every 6 weeks, for up to 17 cycles (approximately 2 years)
  Interventions: Drug: Sitravatinib; Drug: tislelizumab-matching placebo
- Treatment Arm D: Matching Placebo (Experimental): sitravatinib-matching placebo once daily and tislelizumab-matching placebo once every 6 weeks, for up to 17 cycles (approximately 2 years)
  Interventions: Drug: sitravatinib-matching placebo; Drug: tislelizumab-matching placebo

INTERVENTIONS:
Drug: Sitravatinib — Administered orally
  Arms: Treatment Arm A: sitravatinib + tislelizumab; Treatment Arm C:Sitravatinib + Placebo
Drug: Tislelizumab — Administered intravenously
  Arms: Treatment Arm A: sitravatinib + tislelizumab; Treatment Arm B: Placebo + tislelizumab
Drug: sitravatinib-matching placebo — administered orally
  Arms: Treatment Arm B: Placebo + tislelizumab; Treatment Arm D: Matching Placebo
Drug: tislelizumab-matching placebo — administered intravenously
  Arms: Treatment Arm C:Sitravatinib + Placebo; Treatment Arm D: Matching Placebo

SUMMARY:
The purpose of this study is to compare the efficacy and safety of sitravatinib plus tislelizumab or placebo plus tislelizumab versus placebo. The study will also compare the recurrence-free survival (RFS) in participants with hepatocellular carcinoma (HCC) who are at high risk of recurrence after surgical resection.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participant with a first diagnosis of HCC must have undergone a curative-intent resection within 4 to 12 weeks before randomization and have a documented histological confirmation of HCC diagnosis and negative surgical margins (R0 resection) of the resected tumor
2. Participant must have tumor-free status as assessed by the investigator and have fully recovered from surgical resection before randomization
3. Participant must have no extrahepatic HCC
4. ECOG Performance Status ≤ 1
5. Participant who has undergone surgical resection and is defined as having a high risk of HCC recurrence

Key Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC histology
2. Evidence of residual, recurrent, or metastatic disease of HCC before randomization
3. Major macrovascular (gross vascular) invasion of the portal vein (Vp3 or Vp4) or any grade of macrovascular invasion in the hepatic vein or inferior vena cava
4. Untreated chronic hepatitis B (HBV) or chronic HBV carriers with HBV DNA ≥ 2000 IU/mL at Screening
5. Untreated or incompletely treated esophageal or gastric varices with bleeding or high risk of bleeding

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) as assessed by the investigator between Arm A and Arm D | Up to 2 Years
  RFS is defined as the time from the date of randomization until the date of the first documented occurrence of intrahepatic or extrahepatic hepatocellular carcinoma (HCC) as assessed by the investigator, or death from any cause, whichever occurs first.
Recurrence-free survival (RFS) as assessed by the investigator between Arm B and Arm D | Up to 2 Years
  defined as the time from the date of randomization until the date of the first documented occurrence of intrahepatic or extrahepatic hepatocellular carcinoma as assessed by the investigator, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Arm A and Arm B: Recurrence-free survival (RFS) | Up to 2 Years
  defined as the time from the date of randomization until the date of the first documented occurrence of intrahepatic or extrahepatic hepatocellular carcinoma as assessed by the investigator, or death from any cause, whichever occurs first.
Arm A and Arm C: Recurrence-free survival (RFS) | Up to 2 Years
  defined as the time from the date of randomization until the date of the first documented occurrence of intrahepatic or extrahepatic hepatocellular carcinoma as assessed by the investigator, or death from any cause, whichever occurs first.
Arm A and Arm D: overall survival (OS) | Up to 5 Years
  defined as the time from the date of randomization until the date of death due to any cause
Arm B and Arm D: overall survival (OS) | Up to 5 Years
  defined as the time from the date of randomization until the date of death due to any cause
Arm A and Arm B: overall survival (OS) | Up to 5 Years
  defined as the time from the date of randomization until the date of death due to any cause
Arm A and Arm C: overall survival (OS) | Up to 5 Years
  defined as the time from the date of randomization until the date of death due to any cause
Arm A and Arm D: time to extrahepatic spread (EHS) as assessed by the investigator | Up to 2 Years
  defined as the time from the date of randomization until the date of the first documented occurrence of extrahepatic HCC
Arm B and Arm D: time to extrahepatic spread (EHS) as assessed by the investigator | Up to 2 Years
  defined as the time from the date of randomization until the date of the first documented occurrence of extrahepatic HCC
Arm A and Arm B: time to extrahepatic spread (EHS) as assessed by the investigator | Up to 2 Years
  defined as the time from the date of randomization until the date of the first documented occurrence of extrahepatic HCC
Arm A and Arm C: time to extrahepatic spread (EHS) as assessed by the investigator | Up to 2 Years
  defined as the time from the date of randomization until the date of the first documented occurrence of extrahepatic HCC
Number of participants with adverse events (AEs) | Up to 5 Years
  Incidence and severity of adverse events, with severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version (v) 5.0, vital signs, and clinical laboratory test results in the Safety Analysis Set
Participants Reported Outcome as measured at Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) and its hepatocellular carcinoma cancer module QLQ-HCC18 | Up to 2 Years
  Quality of Life change with treatment. Scale scores are calculated by averaging items within scales and transforming average scores linearly. All of the scales range in score from 0 to 100

IPD SHARING:
Plan to Share IPD: Yes